CLINICAL TRIAL: NCT06799247
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial of Descartes-08 in Patients With Generalized Myasthenia Gravis (MG)
Brief Title: Investigating an mRNA CAR T-cell Therapy, Known as Descartes-08, as a Potential Approach to Treat Myasthenia Gravis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNAC-MG-002 (AURORA)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Myasthaenia Gravis
Keywords: myasthenia gravis; CAR-T therapy; Cell Therapy; Decartes-8; BMCA; B cell maturation antigen
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, multi-center phase 3 trial to evaluate the efficacy, safety and tolerability of autologous T-cells expressing a chimeric antigen receptor (CAR) directed to B-Cell maturation antigen (BCMA) in patients with antibody positive gMG. The cell product will be referred to as "Descartes-08".
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: first part of the study is double blinided and the second part of the study is open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decartes-08 (Experimental): This group will undergo leukapheresis and receive manufactured Decartes-08
  Interventions: Biological: Decartes-08
- Placebo (Placebo Comparator): This group will receive placebo
  Interventions: Other: Placebo Drug

INTERVENTIONS:
Biological: Decartes-08 — Autologous mRNA CAR T-cell therapy
  Arms: Decartes-08
Other: Placebo Drug — infusion without Decartes-08
  Arms: Placebo

SUMMARY:
The AURORA Study is evaluating the safety, tolerability, and efficacy of an investigational mRNA CAR T-cell therapy known as Descartes-08 in adults with acetylcholine receptor autoantibody -positive generalized myasthenia gravis. Part 1 of the study will last around 6 months. For eligible participants, Part 2 will last around 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age.
* Patient must have generalized myasthenia gravis (gMG), Myasthenia Gravis Foundation of America (MGFA) clinical classification grades 2-4 at the time of Sscreening.
* MG-Activities of Daily Living (MG ADL) total score ≥ 6.
* Concomitant immunosuppressive drugs must be deemed necessary by the investigator. The dose must be stable for a minimum of 8 weeks prior to Baseline visit.
* If a patient is using corticosteroids, the daily dose should not exceed 40 mg/day of prednisone equivalent. The dose must have been stable for a minimum of 8 weeks prior to Baseline visit.
* Acetylcholine receptor autoantibody (anti-nAChR) titer or anti-AChR cluster antibody must be above the reference laboratory upper normal limit (UNL) and documented within the past 10 years of screening.
* Patient must be willing to return for all study visits.
* Patient must be able to give written informed consent.
* Women of childbearing potential must agree to use highly effective birth control from Screening until 14 days post last dose of Descartes-08,

Exclusion Criteria:

* Major chronic illness that is not well managed at the time of study entry and in the opinion of the investigator may increase the risk to the patient.
* Diagnosis of gMG within 12 months of screening.
* No history of systemic treatment for gMG other than acetylcholine esterase inhibitors.
* Diagnosis of a neuromuscular disease other than gMG.
* Patient is pregnant or lactating.
* Treatment with intravenous immunoglobulin (IVIG) or plasma exchange within 4 weeks prior to the Baseline visit.
* Treatment with rituximab or ocrelizumab within 12 months prior to Baseline visit; treatment with calcineurin inhibitors (e.g. tacrolimus, cyclosporine, cyclophosphamide), Neonatal Fc receptor antagonists, and/or other biologics within 3 weeks prior to planned leukapheresis and within 8 weeks prior to Baseline visit.
* The patient has started treatment with a complement 5a (C5a) inhibitor, such as eculizumab, within 8 weeks of Baseline visit. (NOTE: patients who have been receiving a C5a inhibitor for more than 8 weeks and meet other criteria for enrollment are eligible for treatment).
* Prior treatment with B-cell maturation antigen (BCMA)-directed therapy (e.g. monoclonal antibody, T-cell engager, or chimeric antigen receptor T-cell [CAR-T]).
* Abnormal prothrombin (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) increased > 1.5-fold above the normal range at Screening or patient is on anticoagulation therapy (except in cases of elevated PTT with documented lupus anticoagulant; or in patients who have been on stable doses of anticoagulation therapy for more than 6 months of venous thromboembolism (VTE) diagnosis; or in patients on stable doses of anticoagulation therapy for at least 8 weeks of atrial fibrillation diagnosis; these conditions will not be exclusionary unless, in the investigator's opinion, they make participation in the study unsafe).
* Absolute neutrophil count (ANC) < 1000 cells/microliter.
* Hemoglobin < 8.0 g/dL.
* Platelets < 50,000/mm3.
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3x above normal.
* Creatine clearance less than 30 mL/min.
* History of primary immunodeficiency, organ, or allogeneic bone marrow transplant.
* Patients must be seronegative for hepatitis B surface antigen.
* Patients must be seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patients must be tested for the presence of viremia by reverse transcriptase polymerase chain reaction (RT-PCR) and must be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
* History of positive human immunodeficiency virus (HIV) or positive HIV at screening.
* Active tuberculosis or positive QuantiFERON test at screening.
* Any other clinical or laboratory abnormality that, in the opinion of the investigator, may jeopardize the subject's ability to participate in the study or could affect study outcome.
* Any active significant cardiac or pulmonary disease that, in the opinion of the Principal Investigator, is significant and/or uncontrolled.

Note: Patients with asthma and chronic obstructive pulmonary disease (COPD) controlled with inhaled medications are allowed.

* History of malignancy that required treatment in the past 3 years, except for squamous cell carcinoma, basal cell carcinoma of the skin, or breast or early-stage colon cancer that is surgically removed and did not require adjuvant chemotherapy or radiotherapy.
* Treatment with any investigational agent 4 weeks prior to screening or 5 half-lives of the investigational drug (whichever is longer).
* Receipt of a live vaccination within 4 weeks prior to Baseline visit or intent to receive live vaccination during the study (Note: messenger RNA [mRNA]-based vaccines such as those against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) are not considered live; likewise, the Janssen Covid-19 vaccine is not live).
* History of significant recurrent infections or any active infection that in the opinion of the Investigator may interfere with the patient's participation in the opinion of the investigator.
* Any known psychiatric illness that in the opinion of the Investigator, may interfere with the patient's participation in the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Myasthenia Gravis Activities of Daily Living (MG-ADL) | assessment at 4 months of study
  To evaluate the efficacy of Descartes-08 as assessed by the proportion of Myasthenia Gravis Activities of Daily Living (MG-ADL) responders at Month 4.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (14):
  - A40, Tucson, Arizona
  - A13, Carlsbad, California
  - A14, Orange, California
  - A21, Aurora, Colorado
  - A48, Maitland, Florida
  - A10, Tampa, Florida
  - A53, O'Fallon, Illinois
  - A20, Fairway, Kansas
  - A38, Boston, Massachusetts
  - A12, Amherst, New York
  - A47, New York, New York
  - A22, Chapel Hill, North Carolina
  - A43, Houston, Texas
  - A41, Seattle, Washington
- A23, Rome, Italy
- A30, Krakow, Poland
- A24, Belgrade, Serbia
- Spain (2):
  - A25, Barcelona
  - A31, Madrid
- Turkey (Türkiye) (2):
  - A32, Ankara
  - A17, Istanbul

IPD SHARING:
Plan to Share IPD: No